CLINICAL TRIAL: NCT01780441
Title: Longitudinal Study to Identify Early Biomarkers of Autism Spectrum Disorder (ASD) in Infants With Tuberous Sclerosis Complex (TSC)
Brief Title: Early Biomarkers of Autism in Infants With Tuberous Sclerosis Complex (TSC)
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Tuberous Sclerosis Alliance (Other)
Responsible Party: Principal Investigator, Mustafa Sahin, MD, PhD, Boston Children's Hospital
Other Study IDs: IRB-P00005074; 1U01NS082320-01 (NIH)
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Tuberous Sclerosis Complex; TSC; Autism; ASD; Biomarkers; Infants
MeSH Terms: conditions — Tuberous Sclerosis; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tuberous Sclerosis Complex (TSC): Tuberous Sclerosis Complex

SUMMARY:
The investigators are enrolling 3-12 month old infants with a diagnosis of tuberous sclerosis complex (TSC) for a new study on early markers of autism. The study is looking for early signs for autism in a population (TSC) where autism is common. The goal of this project is to use behavioral testing, MRI and EEG techniques to identify children at risk for developing autism starting at 3 months of age and continuing until 36 months of age. Throughout the study, the investigators will recommend Early Intervention services for any child who shows early signs of autism.

DETAILED DESCRIPTION:
This is a five-year multi-site study using MRI and EEG technologies to identify developmental precursors of Autism Spectrum Disorder in patients with Tuberous Sclerosis Complex (TSC). The study will be enrolling infants at five TSC centers throughout the country, including Boston Children's Hospital, Cincinnati Children's Hospital Medical Center, University of Alabama at Birmingham, University of Texas at Houston and University of California Los Angeles. The main goal of this study is to identify early signs of autism in children with TSC looking at the brain through MRI/diffusion tensor imaging, EEG and behavioral/neuropsychological methods. Eligible infants between the ages of 3-12 months will be evaluated longitudinally at regular visit intervals up to 3 years of age.

Study Objectives

1. To characterize the developmental precursors of ASD in a large number of TSC infants using a prospective multi-center design: Infants with TSC will be evaluated longitudinally at ages 3, 6, 9, 12, 18, 24 and 36 months. At each age, children will undergo standardized evaluations, using cognitive and adaptive measures. At age 24 and 36 months, formal assessment for autism will be performed. Clinical data including medication use, seizure history, EEG activity, genotypic variation, and co-morbidities will be recorded to determine if specific clinical factors modify the course of development.
2. To identify biomarkers with advanced diffusion tensor imaging (DTI) that help predict development of ASD in TSC infants: The investigators hypothesize that decreased white matter integrity performed annually for each of the first 3 years of life, including DTI sequences with tractography. Radial, axial, and mean diffusivity and fractional anisometry will be calculated for each time point and change over time correlated with development of ASD to determine relative risk. Individual measures at each time point will be compared between ASD and non-spectrum groups to assess the individual impact of each measure and timing.
3. To identify biomarkers with quantitative EEG that help predict development of ASD in TSC infants: The investigators hypothesize that altered functional connectivity, as measured by qEEG coherence and high frequency oscillations, will correlate with development of ASD in TSC. Quantitative EEG (qEEG), EEG coherence/gamma frequency (30-50Hz), and high frequency oscillations encompassing both ripples (80-250H) and fast ripples (250-500 Hz) will be measured at each time point. Changes over time will be correlated with development of ASD to determine relative risk, as will comparison of individual measures between the two groups. EEG findings will also be correlated with MR results obtained to further couple functional connectivity as measured by EEG with structural connectivity measured by DTI.

ELIGIBILITY:
Inclusion Criteria:

1. Meets genetic or clinical diagnostic criteria for TSC (Tuberous Sclerosis), the latter based on current recommendations for diagnostic evaluation, such as physical exam, neuroimaging, echocardiogram.
2. Age criteria: 3 months- 12 months of age at time of enrollment. For study purposes, 3 months is defined as ≥ 9 weeks, 1 day and 12 months is defined as ≤ 13.5 months.

Exclusion Criteria:

1. Prematurity, defined as gestational age < 36 weeks at time of delivery
2. Has taken an investigational drug as part of another research study, within 30 days prior to study enrollment
3. Is taking an mTOR inhibitor such as rapamycin, sirolimus, or everolimus (other than topical formulations) at the time of study enrollment
4. Subependymal Giant Cell Astrocytoma requiring medical or surgical treatment at the time of study enrollment
5. History of epilepsy surgery at the time of study enrollment
6. Contraindications to MRI scanning, such as metal implants/non-compatible medical devices or medical conditions

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 150 evaluable infants with TSC will be recruited. Diagnosis of TSC will be based on established clinical criteria and will not require genetic testing prior to participation. The target age of entry into study is 3-6 months, but infants up to age 12 months (less than or equal to 13.5 months) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
ADOS evaluation score at the 36 month visit | 36 months
  The ADOS performed at 24 and 36 months will be used as a preliminary diagnosis for data analysis. The primary outcome is the possible clinical diagnosis of autism spectrum disorder per the DSM 5 guidelines (Autistic Disorder, Asperger's and PDD-NOS).
MRI biomarkers | 36 months
  MRI biomarkers obtained at baseline, 12, 24, 36 months will be applied to characterize individual patients in terms of brain tissue, white matter structure and connectivity, functional networks, and pathology. Brain tissue segmentation will be based on structural images derived from T1- and T2-weighted and FLAIR sequences using automated software tools designed for these tasks. White matter integrity and organization will be inferred from DTI imaging sequences. Structural connectivity networks will be delineated by DTI tractography assessment.
EEG biomarkers | 36 months
  One-hour video-EEG containing both wakefulness and sleep (minimum of 20 minutes of each) will be obtained at baseline, 3, 6, 9, 12, 18, 24 and 36 months. Functional connectivity and pathological activity will be determined by measurement of EEG coherence and gamma frequency/high frequency oscillations.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Sahin, MD, PhD, Principal Investigator — Boston Children's Hospital; Darcy Krueger, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at Los Angeles, Los Angeles, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas at Houston, Houston, Texas

REFERENCES:
- [Derived] Srivastava S, Prohl AK, Scherrer B, Kapur K, Krueger DA, Warfield SK, Sahin M; TACERN Study Group. Cerebellar volume as an imaging marker of development in infants with tuberous sclerosis complex. Neurology. 2018 Apr 24;90(17):e1493-e1500. doi: 10.1212/WNL.0000000000005352. Epub 2018 Mar 23. PMID 29572283
- See also: Boston Children's Hospital - Multi-Disciplinary Tuberous Sclerosis Program — http://www.tsclinic.org/
- See also: Tuberous Sclerosis Alliance — http://www.tsalliance.org/
- See also: TSC Clinic at Cincinnati Children's Hospital Medical Center — http://www.cincinnatichildrens.org/service/t/tuberous-sclerosis/default/
- See also: Study website — http://www.tscstudy.com/